CLINICAL TRIAL: NCT01039558
Title: Randomized Controlled Trial to Evaluate the Effect of Lansoprazole in Combination With Ecabet Sodium for Gastroesophageal Reflux Disease
Brief Title: The Effect of Lansoprazole in Combination With Ecabet Sodium for Gastroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Joo Sung Kim, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RECURRENT GERD
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: gastroesophageal reflux disease; lansoprazole; ecabet sodium
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — ecabet; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lansoprazole + ecabet sodium (Active Comparator)
  Interventions: Drug: ecabet sodium; Drug: lansoprazole
- lansoprazole + placebo (Placebo Comparator)
  Interventions: Drug: lansoprazole; Drug: placebo

INTERVENTIONS:
Drug: ecabet sodium — Active comparator group patients will take lansoprazole 15 mg once daily and ecabet sodium 1.0 g three times daily and placebo group patients will take lansoprazole 15 mg once daily and placebo 1.0 g three times daily for total 8 weeks.
  Other Names: Gastrex ganules
  Arms: lansoprazole + ecabet sodium
Drug: lansoprazole — Active comparator group patients will take lansoprazole 15 mg once daily and ecabet sodium 1.0 g three times daily and placebo group patients will take lansoprazole 15 mg once daily and placebo 1.0 g three times daily for total 8 weeks.
Drug: placebo — Active comparator group patients will take lansoprazole 15 mg once daily and ecabet sodium 1.0 g three times daily and placebo group patients will take lansoprazole 15 mg once daily and placebo 1.0 g three times daily for total 8 weeks.
  Arms: lansoprazole + placebo

SUMMARY:
We will estimate the responses of lansoprazole and ecabet sodium combination therapy and compare with lansoprazole and placebo therapy in patients who need additional therapy after standard proton pump inhibitor treatment for 4week or more in recurrent gastroesophageal reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* age 19-75 years
* patients with typical gastroesophageal symptom or erosive reflux esophagitis on gastroduodenoscopy
* patients with recurrent gastroesophageal symptom after standard proton pump inhibitor treatment for 4 weeks or more

Exclusion Criteria:

* patients with gastric ulcer or duodenal ulcer
* patients with gastric cancer or esophageal cancer
* pregnant or postpartum women

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
We will compare the summations of symptoms score and calculate the response rate | after 4 weeks and 8 weeks

SECONDARY OUTCOMES:
the global response of treatment | after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joo Sung Kim, M.D., PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea